CLINICAL TRIAL: NCT06002113
Title: Assessment of Shared Decision-making Tool for Eliciting Informed Goals of Care in the Hospitalized Elderly (ASKMEGOC): A Randomized Clinical Trial
Brief Title: Eliciting Informed Goals of Care in Elderly Patients
Acronym: ASKMEGOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Victoria Hospital, Canada (Other)
Collaborators: Royal Victoria Regional Health Centre (Unknown)
Responsible Party: Principal Investigator, Giulio DiDiodato, Chief Research Scientist, Royal Victoria Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R22-003
Record Dates: First submitted 2023-07-27; First posted 2023-08-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Goals of Care; Patient Preference; End of Life
MeSH Terms: conditions — Patient Preference; Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOCD Tool (Experimental): Intensive care unit-facilitated goals-of-care discussion using web-based shared-decision making software tool
  Interventions: Other: GOCD Tool
- usual care (Active Comparator): Usual discussions conducted by attending physician with patient
  Interventions: Other: Usual care

INTERVENTIONS:
Other: GOCD Tool — Web-based tool with 4 components; pre-admission health status; current illness prognosis for hospital survival; in-hospital cardiorespiratory arrest prognosis; values and goals of care
  Arms: GOCD Tool
Other: Usual care — Attending physicians responsible for GOCD during hospitalization using their usual approaches
  Arms: usual care

SUMMARY:
Patient-centered medical care considers a patient's values and goals for their health and well-being. Healthcare providers use this information to formulate a medical care plan that is aligned with these expectations. This shared-decision making process should occur with every medical decision, but it is especially important whenever decisions about end-of-life care are being considered. Eliciting patient preferences about resuscitation and life-support treatments in the event of life-threatening illnesses are considered to be a standard of excellent and appropriate medical care. Unfortunately, these discussions don't happen consistently and even when they do occur, are rarely ideal. The consequences can be devastating, often resulting in the delivery of unwanted medical care that can be associated with significant physical and mental suffering among patients and their families. In response to this problem, the investigators developed a novel tool to help guide these difficult conversations between healthcare providers and patients. The investigators previously tested this tool in a small group of hospitalized patients who found it acceptable and helpful. In this larger study, the investigators will compare how effective this tool is compared to usual care in ensuring hospitalized patients have their treatment preferences identified, documented and result in end-of-life care that is consistent with their preferences.

DETAILED DESCRIPTION:
Objectives:

1. To determine the impact of facilitated Goals of Care Discussions (GOCDs) on the number of ICU, ventilator, and dialysis days during the index hospitalization (or until death) (composite).
2. To determine the impact of facilitated GOCDs on the number of ICU, ventilator, and dialysis days after the index hospitalization until 12 months post-admission from the index hospitalization (or until death) (composite).
3. To determine the impact of f-GOCDs on the final treatment preferences for life sustaining treatments (LSTs) documented in CODE STATUS.
4. To determine the impact of facilitated GOCDs on other outcomes including decisional conflict and quality of communication, patient satisfaction with the encounter, and place of death.
5. To determine the difference in direct patient hospital costs
6. To determine the barriers and facilitators to the implementation of GOCDs.

Design:

A prospective, single-centre, stratified, parallel group, allocation concealed, analyst-masked, randomized, pragmatic, mixed-method, comparative effectiveness trial in hospitalized elderly patients 80 years and older.

Participants:

This study will include all elderly patients admitted to the Royal Victoria Regional Health Centre in Barrie, Ontario, Canada, with an acute medical or surgical diagnosis who fulfill all the inclusion criteria and for whom none of the exclusion criteria exist.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients ≥ 80 years old with an acute medical or surgical condition admitted to any hospital ward
* Previously or currently documented CODE STATUS preferences include any life sustaining therapies
* Duration of admission ≥ 24 hours
* English speaking, or translator present
* Competent patient or substitute decision maker

Exclusion Criteria:

* Treating physician, patient, or substitute decision maker declines
* Documented resuscitation preferences for comfort or supportive care
* New diagnosis of life-limiting illness on this hospital admission, for example, new diagnosis of metastatic cancer
* Clinically unstable, admitted to an intensive care unit, or currently receiving acute life support treatment (mechanical ventilation, acute dialysis, or inotropic/vasopressor support)
* Readmission after index hospitalization
* Pre-existing need for chronic mechanical ventilation (invasive mechanical ventilation via tracheostomy > 90 days) or maintenance dialysis (peritoneal or hemodialysis > 90 days)

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
ICU-related health care utilization | From the time of index hospital admission until hospital discharge or death, up to 12 months after the time of index hospital admission
  total number of ventilator, ICU, and dialysis days
ICU-related health care utilization | 12 months after admission from index hospital admission
  total number of hospital, ventilator, ICU, and dialysis days

SECONDARY OUTCOMES:
CODE STATUS resuscitation preferences | At the time of index hospital discharge or death during the index hospitalization, up to 12 months after the time of index hospital admission
  Distribution of resuscitation preferences documented in CODE STATUS
Change in CODE STATUS preferences | At the time of index hospital discharge or death during the index hospitalization, up to 12 months after the time of index hospital admission
  Proportion of patients who change documented CODE STATUS preferences
Resuscitation level designation | At the time of index hospital discharge or death, up to 12 months after the time of index hospital admission
  proportion of patients with completed resuscitation preferences identified
Distribution of ICU-related days of health care utilization | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  compare empirical distributions of total days of health care utilization
Time required to complete GOCD-facilitated discussion | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  Total time required to complete intervention
Quality of communication | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  assessment of patient perceptions of quality of goals of care discussion
patient satisfaction with GOCD discussion | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  patient satisfaction with goals of care discussions
Evaluation of GOCD tool | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  patient's perceptions of quality of web-based tool
Patient-provider agreement on resuscitation preferences | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  decision concordance between patients and providers
Death | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  date and time and place of death during study period
Direct hospital costs | From index hospital admission until hospital discharge or death in hospital, assessed up to 12 months
  Difference in direct hospital costs

CONTACTS AND LOCATIONS:
Overall Officials: Giulio DiDiodato, MD PhD, Principal Investigator — Royal Victoria Regional Health Centre; Chris Martin, MD, Principal Investigator — Royal Victoria Regional Health Centre; Doug Austgarden, MD, Principal Investigator — Royal Victoria Regional Health Centre
Locations (1):
- Royal Victoria Regional Health Centre, Barrie, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only upon request, de-identified data may be shared

REFERENCES:
- [Derived] Martin C, Cruise K, Aggarwal M, Austgarden D, DiDiodato G. Assessment of shared decision-making tool for eliciting informed goals of care in the hospitalized elderly (ASKmeGOC): protocol for a randomized clinical trial. Trials. 2025 Dec 16. doi: 10.1186/s13063-025-09323-6. Online ahead of print. PMID 41402864